CLINICAL TRIAL: NCT06993896
Title: Assessment of Physical Activity During Chemo- and/or Immunotherapy for Lung Cancer
Brief Title: Physical Activity During Chemo- and/or Immunotherapy for Lung Cancer
Acronym: APACHIE-01
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Other Study IDs: APACHIE-01
Record Dates: First submitted 2025-05-16; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer (NSCLC)
Keywords: lung cancer; chemotherapy; immunotherapy; physical activity
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with steps counted by their smart phone: The purpose is to obtain a patient's mean number of steps per week directly from the patient's smart phone which has a step counter.

SUMMARY:
The main goal of this trial is to describe the pattern of physical activity in patients with non-small cell lung cancer during chemo- and/or immunotherapy, to evaluate potential predictors of those patterns and to assess potential correlations with patient reported outcomes (pain-, distress-, and fatigue scores). To reach this goal, this trial will be first trial in which the mean number of steps per week performed at baseline and during each week of chemo- and or immunotherapy will be collected in a standardized prospective way. The trial is exploratory in nature with the aim to generate scientific hypotheses to be investigated in future clinical trials.

DETAILED DESCRIPTION:
Lung cancer belongs to the most common types of solid cancer in Europe and Northern America. Most patients with non-small cell lung cancer receive chemo- and/or immunotherapy. Many patients with distant metastases (stage IV disease) are treated with chemo- and/or immunotherapy alone or combined with palliative radiotherapy. Moreover, a considerable number of patients assigned to thoracic surgery receive neoadjuvant chemo- and/or immunotherapy without irradiation. The chemo- and/or immunotherapy regimens used for non-small cell lung cancer may be associated with adverse events including fatigue. Patients who experience significant treatment-related toxicity may not be able to receive the complete chemo- and/or immunotherapy as planned. Physical activity may be helpful in this context. In a retrospective study, adherence to an exercise program was associated with fewer dose reductions and delays of chemotherapy. Moreover, several studies performed in patients with lung cancer suggested that physical activity had a positive effect on the patient's quality of live. Thus, physical activity prior to and during chemo- and/or immunotherapy for lung cancer appears important.

Adherence to an exercise program sometimes may be challenging for the patients, particularly if they experience treatment-related fatigue or other adverse events. The question arose whether an easy-to-use mobile app installed on the patient's smart phone reminding patients several times daily to perform a certain number of steps will have a positive effect on their physical activity during chemo- and/or immunotherapy. The patient's smart phone will also be used for counting the steps. Such an app is currently under development within the European Territorial Co-Operation project "Health Advancing Technologies for Elderly (HeAT)". This app will be tested in a prospective phase 2 trial. For proper sample size calculation and design of the trial, the current prospective study is required, which evaluates the weeks with a mean number of steps per week at baseline and during chemo- and/or immunotherapy for non-small cell lung cancer.

The main goal of this trial is to evaluate patterns and predictors of physical activity during chemo- and/or immunotherapy for lung cancer. The primary endpoint is to assess the mean number of steps per week during the first three cycles of chemo- and/or immunotherapy for lung cancer. The baseline value is represented by the mean number of steps during the last week prior to chemotherapy and/or immunotherapy. Any type of smart phone is allowed, as long as it has a step counter. In addition, associations between mean number of steps per week and a pain-score, a distress-score and a fatigue-score will be evaluated. The recruitment of all 38 patients should be completed within 4 months. The treatment period will be 9-10 weeks (three cycles of chemo- and/or immunotherapy). This equals a total running time for the trial of approximately 6 months.

Sample size calculation: Due to the exploratory character of this trial, sample size estimation is not based on a specific statistical hypothesis system. Instead, the sample size is derived by the following simple statistical reasoning and feasibility aspects. The goal of this study is to compare mean number of steps per week between various study weeks. Therefore, the effect size is considered as a relevant parametrization of the shift in mean values. The effect size defined as the mean of the paired difference divided by its standard deviation, and therefore, constitutes a standardized scale indicating the number of standard deviations by which the means differ. Assuming that an effect size of 0.5 for the mean number of steps per week between two study weeks is clinically interesting/relevant and worth to be detected, 34 patients are required to achieve a power of 80% with a level of significance of 5% (two-sided) using a t-test for comparing two paired means. This sample size is also considered feasible in this single-center trial setting considering the planned study duration. Assuming that 10% of the patients may not be included in the descriptive analyses due to lack of data, a total number of 38 patients should be enrolled to this exploratory, hypothesis-generating trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven non-small cell lung cancer
2. Indication for chemo- and/or immunotherapy
3. Possession of and ability to use a smart phone that includes a step counter
4. Willingness to wear the smart phone close to the body at any time
5. Age ≥18 years
6. Written informed consent
7. Capacity of the patient to consent

Exclusion Criteria:

1. Small-cell lung cancer
2. Karnofsky performance score <60
3. Thoracic surgery within 3 months prior to chemo- and/or immunotherapy
4. Expected Non-Compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy and/or immunotherapy for non-small cell lung cancer who possess a smart phone with a step counter.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean number of steps per week performed at baseline and during the first three cycles of chemo- and/or immunotherapy for lung cancer | through study completion, 9 weeks
  The primary endpoint is to assess the mean number of steps per week during the first three cycles of chemo- and/or immunotherapy for lung cancer. The baseline value is represented by the mean number of steps during the last week prior to chemotherapy and/or immunotherapy. Any type of smart phone is allowed, as long as it has a step counter.

SECONDARY OUTCOMES:
Degree of the impact of pain on the mean number of steps per week asessed using the Numeric Pain Rating Scale | through study completion, 9 weeks
  Pain will be assessed prior to chemo- and/or immunotherapy, weekly during the three cycles of chemo- and/or immunotherapy, and at end of treatment with the Numeric Pain Rating Scale (self-assessment, ranging from 0 points = no pain to 10 points = maximum pain). Pain scores of 0-5 points will be compared to pain scores of 6-10 points.
Degree of the impact of distress on the mean number of steps per week asessed using the Distress Thermometer | through study completion, 9 weeks
  Distress will be assessed prior to chemo- and/or immunotherapy, weekly during the three cycles of chemo- and/or immunotherapy, and at end of treatment with the Distress Thermometer (self-assessment, ranging from 0 points = no distress to 10 points = maximum distress). Distress scores of 0-5 points will be compared to distress scores of 6-10 points.
Degree of the impact of fatigue on the mean number of steps per week asessed using the Fatigue Asessment Scale (FAS) | through study completion, 9 weeks
  Fatigue will be assessed prior to chemo- and/or immunotherapy, weekly during the three cycles of chemo- and/or immunotherapy, and at end of treatment with the Fatigue Assessment Scale (FAS) (self-assessment, ranging from 0 points = no fatigue to 50 points = maximum fatigue) [© FAS (Fatigue Assessment Scale)]. Fatigue scores of 0-21 points (no fatigue) will be compared to fatigue scores of 22-50 points (substantial fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr. med., Principal Investigator — University of Lubeck

IPD SHARING:
Plan to Share IPD: No